CLINICAL TRIAL: NCT04503408
Title: A Comparison of Pulmonary Function, Functional Capacity, Muscle Strength, Physical Activity, Physical Fitness and Activities of Daily Living in Cystic Fibrosis Patient's With and Without Abnormal Glucose Tolerance.
Brief Title: A Comparison of Clinical Parameters in With and Without Abnormal Glucose Tolerance.
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Kocaaga, Principal investigator, Hacettepe University
Other Study IDs: GO19/704
Record Dates: First submitted 2020-04-07; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Cystic Fibrosis-related Diabetes; Diabetes Mellitus; Cystic Fibrosis
Keywords: Glucose; Cystic fibrosis; Muscle strength; Physical fitness
MeSH Terms: conditions — Diabetes Mellitus; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cystic fibrosis with abnormal glucose tolerance: cystic fibrosis with abnormal glucose tolerance Cystic fibrosis patients with descripted that impaired glucose tolerance or cystic fibrosis related diabetes by oral glucose tolerance test
- cystic fibrosis with normal glucose tolerance: cystic fibrosis with normal glucose tolerance Cystic fibrosis patients with descripted that normal glucose tolerance by oral glucose tolerance test

SUMMARY:
Cystic fibrosis (CF) is autosomal recessive, genetic disorder cause of cystic fibrosis transmembrane regulatory (CFTR) gene mutation. CF often is observed in caucasian population. CFTR protein in cell apical membrane is canal responsible of transport sodium and clorid ions. Impaired sodium ion transport causes production viscous mucus. Disease include problems such as mucus, breathlessness and coughing. Blood glucose levels fluctuation are observed. This study aims comparison between lung function, functional capacity, muscle strength, physical activity, physical fitness and activities of daily living activities in cystic fibrosis with and without abnormal glucose tolerance

DETAILED DESCRIPTION:
The study aimed that comparison of clinical parameters in children with and without abnormal glucose tolerance in Cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Cystic fibrosis with impaired glucose tolerance or cystic fibrosis-related diabetes for Abnormal glucose tolerance group
2. Cooperation for tests
3. Indıviduals without an orthopedic or neurological problem and serious cardiac problems that effecting tests,
4. To volunteer for the study.

For the control group

1. Cystic fibrosis with normal glucose tolerance
2. Cooperation for tests
3. Indıviduals without an orthopedic or neurological problem and serious cardiac problems that effecting tests,
4. To volunteer for the study.

Exclusion Criteria:

Patients having following disease

1. Acute pulmonary exacerbation
2. Acute or chronic respiratory failure
3. FEV₁ lower than %40
4. Cooperation problems,
5. Bronchopulmonary aspergillus and using steroid.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: cystic fibrosis with (impaired glucose tolerance, cystic fibrosis related diabetes) and without abnormal glucose tolerance
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Distance of 6 minute walk test | 28 week
  Distance of 6 minute walk test assesing functional capacity made on flat corridor with speed is determined from participant. She/he walks during 6 minute on this corridor as quickly as possible.
Lung function | 28 week
  Lung function will be assesed for standardization procedure in Cystic fibrosis. Acceptible outcome will be recorded.
Respiratory muscle strength | 28 week
  Both inspiratory and expiratory muscle strength wil be evaluated at least three times in Cystic fibrosis. Mouth pressure device will be used for evaluate. The highest value for MIP and MEP will be recorded.
Quadriceps muscle strength | 28 week
  Quadriceps muscle strength will be assessed least three times in children with cystic fibrosis. hand held dynamometer will be used for assessing quadriceps muscle strength. The highest value for each side will be recorded and used for analysis.
Handgrip | 28 week
  Handgrip will be assessed in Cystic fibrosis using hand dynamometer (Jamar hand dynamometer). Assessing will be repeated three times end mean of three measurement will be calculated and used for analysis.
Physical activity levels | 28 week
  Physical activity will be evaluated with Bouchard physical activity record. This activity recorder is evaluated every 15 min in a day. Two weekday and one weekend day are recorded with made activity.
Physical fitness | 28 week
  Physical fitness is measured with Munich physical fitness test battery. This battery vertial jump, bouncing ball, flexibilty, climbing, throwing bag, step up test are included in battery. the battery evaluates such as strength, endurance, speed, flexibilty, coordination, power.
Distance of shuttle walk test | 28 week
  Distance of shuttle walk test will be walked by children with cystic fibrosis. Shuttle walk test is made on floor with ten meters distance. Speed is determined according to signals from CD player.
Time of activities of daily living test | 28 week
  Activities of daily living will be tested with the Glittre ADL test. This test includes five repeated cycles that includes sitting, walk, step up and changing place of object on bookshelf in test procedure. The total completion time of five cycles will be recorded and used for analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Kocaaga, Ankara, Turkey (Türkiye)